CLINICAL TRIAL: NCT00558207
Title: A Randomized Phase 2 Study of ARQ 197 Versus Gemcitabine in Treatment-Naïve Patients With Unresectable Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-205
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic cancer; pancreas cancer; Locally advanced or metastatic pancreatic adenocarcioma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ARQ 197; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ARQ 197
  Interventions: Drug: ARQ 197
- 2 (Active Comparator): Gemcitabine
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: ARQ 197 — 120 mg capsule administered twice daily for 240 mg total daily dose
  Arms: 1
Drug: gemcitabine — 1000 mg/m2 administered as an intravenous infusion over 30 minutes once weekly for 4 weeks for the first 28 days (cycle). Each subsequent cycle will consist of 1000 mg/m2 administered as an intravenous infusion over 30 minutes once weekly for 3 weeks with no drug administered in the 4th week.
  Other Names: Gemzar
  Arms: 2

SUMMARY:
This is a multi-center, open-label randomized phase 2 study designed to assess the progression free survival (PFS) of patients with untreatment and unresectable pancreatic cancer following treatment with either ARQ 197 or gemcitabine. The study will also evaluate other efficacy and safety endpoints including overall response rate, overall survival and adverse events in the two treatment arms.

DETAILED DESCRIPTION:
This is a multi-center, open-label randomized phase 2 study designed to evaluate the PFS of treatment-naïve patients with unresectable (locally advanced or metastatic) pancreatic adenocarcinoma following treatment with either ARQ 197 (ARQ arm) or gemcitabine alone (GEM arm). The study will also evaluate other efficacy and safety parameters including ORR, OS and adverse events in the two treatment arms. Patients randomly assigned to the GEM arm will receive gemcitabine alone. Patients assigned to the ARQ arm will receive oral ARQ 197 alone.

ARQ 197 is an investigational oral drug supplied as capsules in multiple strengths. For the study initial shipment the capsules were 120 mg each, 30 count. In the ARQ arm, patients will take 120 mg of ARQ 197 twice daily, once in the morning and once in the evening one hour prior to or two hours after a meal. ARQ 197 treatment will be continued until unacceptable toxicity, documented progression of disease, or another discontinuation criterion is met.

Gemcitabine is a commercially available drug for the treatment of patients with locally advanced or metastatic adenocarcinoma of the pancreas. In the GEM arm, gemcitabine will be administered by intravenous infusion over 30 minutes at a dose of 1000 mg/m2. The dosing schedule of gemcitabine will be once weekly for the first cycle (4 weeks), then once weekly for 3 consecutive weeks followed by a week of rest for each subsequent cycle. Gemcitabine therapy will be continued until unacceptable toxicity, documented progression of disease, or another discontinuation criterion is met.

A treatment cycle is defined as 28 days for both treatment arms. Cycles may be repeated every 4 weeks (28 days) based on toxicity and response. The assigned treatment should continue until unacceptable toxicity, disease progression (clinical or radiological) or another discontinuation criterion is met.

Tumor evaluations: Tumor evaluations will be performed in 8-week intervals. Tumor response (complete response, partial response, stable disease, progressive disease and ORR) will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST).

Progression-free survival: The time of disease progression-free will be calculated from randomization until disease progression per RECIST or death due to any cause. Patients who are alive and progression free will be censored at the date of their last tumor evaluation.

Overall survival: Overall survival time will be calculated from the date of randomization until death due to any cause.

Safety assessments: Data on vital signs, physical examination, adverse events, serum chemistry, hematological laboratory tests, and electrocardiograms will be collected.

This study is designed to establish potential efficacy of ARQ 197 in treatment naive pancreatic cancer patients in a controlled, randomized study. The sample size of 30 Evaluable patients per treatment group is considered adequate to provide meaningful estimates of the PFS and ORR and OS rates, however, this study is not powered to show statistically significant differences between the treatment groups. Therefore, the analyses will be primarily descriptive in nature. Taking into account an anticipated drop-out/loss-to-follow-up rate of 20%, the total sample size will be 72 patients.

Primary and secondary objectives will be analyzed in the two treatment arms using appropriate patient populations and statistical methods.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated informed consent prior to study-specific screening procedures
2. ≥ 18 years old
3. Histologically or cytologically confirmed locally advanced or metastatic unresectable pancreatic adenocarcinoma
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
5. Karnofsky performance status (KPS) ≥ 70%
6. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment
7. Females of childbearing potential must have a negative serum pregnancy test
8. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 × ULN with metastatic liver disease
9. Hemoglobin ≥ 10 g/dl
10. Total bilirubin ≤ 1.5 × ULN
11. Serum creatinine ≤ 1.5 x ULN
12. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
13. Platelets ≥ 100 x 10^9/L

Exclusion Criteria:

1. Received any prior therapy for the treatment of their pancreatic malignancy (including chemotherapy, immunotherapy, vaccines, monoclonal antibodies, major surgery, or irradiation, whether conventional or investigational)
2. Central nervous system metastases
3. Pregnant or breastfeeding
4. Significant gastrointestinal disorder, in the opinion of the Principal Investigator (e.g. Crohn's disease, ulcerative colitis, extensive gastric resection)
5. Unable or unwilling to swallow ARQ 197 capsules twice daily
6. Other cancer within the last five years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin
7. Significant co-morbid conditions that in the opinion of the Investigator would impair study participation
8. Known human immunodeficiency virus (HIV) or hepatitis C virus (HCV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Evaluate progression-free survival (PFS) in patients receiving ARQ 197 versus gemcitabine. | 6 month

SECONDARY OUTCOMES:
Evaluate overall response rate (ORR) in patients receiving ARQ 197 versus gemcitabine | ongoing
Evaluate 6-month and 1-year overall survival (OS) rates in patients treated with ARQ197 versus gemcitabine | 6 and 12 month
Further characterize the safety profile of ARQ 197 | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Cezary Szczylik, PhD, Principal Investigator — Klinika Onkologii WIM; Janusz Pawlega, PhD, Principal Investigator — Oddzial Kliniczny Kliniki Onkologii; Piotr Koralewski, MD, Principal Investigator — Oddzial Chemioterapii Krakow; Emilia Filipczyk-Cisarz, MD, Principal Investigator — Oddzial Chemioterapii Dolnoslaskie Centrum Onkologii; Ewa Kilar, MD, Principal Investigator — Regionalny Szpital Specjalistyczny Latawiec; Piotr Sawrycki, MD, Principal Investigator — Oddzial Onkologii Klinicznej im L Rydygiera
Locations (6):
- Poland (6):
  - Oddzial Kliniczny Kliniki Onkologii Szpital Uniwersytecki w Krakowie, Krakow
  - Oddzial Chemioterapii, Wojewodzki Szpital Specjalistyczny, Krakow
  - Oddział Onkologii Klinicznej, Regionalny Szpital Specjalistyczny "Latawiec", Swidnica
  - Oddział Onkologii Klinicznej SP ZOZ Wojewódzki Szpital Zespolony im. L. Rydygiera, Torun
  - Klinika Onkologii WIM Warszawa, Warsaw
  - Oddział Chemioterapii Dolnośląskie Centrum Onkologii, Wroclaw